CLINICAL TRIAL: NCT06833879
Title: A Pilot Study to Evaluate the Use of a Wrist-worn Accelerometer Device for Physical Activity Monitoring in Healthy Volunteers
Brief Title: Activity Tracking Study in Healthy Volunteers (MK-0000-419)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0000-419; MK-0000-419 (Other: MSD)
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Watch Wearing to Track Activity (Experimental): Participants wear a watch that tracks physical activity throughout study.
  Interventions: Device: Activity Tracking Watch

INTERVENTIONS:
Device: Activity Tracking Watch — Device includes a wristwatch that tracks physical activity and a data storage unit that transmits data to a central database.
  Other Names: CentrePoint Insight Watch (ActiGraph) and Data Hub

SUMMARY:
In this study, researchers want to learn if a watch can be used to track physical activity in healthy people. The watch will collect the data and send it to a database using a data storage device.

The goal of this study is to measure:

* The number of people who wear the watch as instructed
* The number of working watches and data storage devices returned at the end of the study
* The number of watches that successfully sent data back to a database
* The overall daily activity for people including the number of daily steps taken and how much time is spent doing non-exercise activity and mild to intense exercise.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to:

* Is in good health
* Is willing to comply with study restrictions

Exclusion Criteria:

The key exclusion criteria include but are not limited to:

* History of clinically significant endocrine, GI, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* History of cancer

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants that Wear Watch as Instructed | Up to approximately 2 weeks
  The number of participants that wear the watch for at least 19.2 hours per day (80% of the time) will be reported.
Number of Provisioned Watches and Data Storage Devices That Were Returned | Up to approximately 2 weeks
  The number of watches and data storage devices provisioned and returned free from malfunction will be reported.
Number of Watches and Data Storage Devices that Successfully Transmit Data | Up to approximately 2 weeks
  The number of watches and data storage devices that successfully transmit data to central database will be reported.
Average Daily Overall Activity Count | Up to approximately 2 weeks
  The average daily overall activity will be reported.
Average Daily Total Step Count | Up to approximately 2 weeks
  The number of average daily total steps will be reported.
Average Daily Time (minutes) in Nonsedentary Activity | Up to approximately 2 weeks
  The average daily time spent in nonsedentary activity will be reported.
Average Daily Time (minutes) in Moderate-to-Vigorous Physical Activity | Up to approximately 2 weeks
  The average daily time spent in moderate-to-vigorous physical activity will be reported.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 2 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 2 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  The number of participants who discontinue study intervention due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - QPS-MRA, LLC (Site 0001), South Miami, Florida
  - Altasciences Clinical Kansas, Inc. (Site 0002), Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com